CLINICAL TRIAL: NCT06911242
Title: A Comparative, Randomized, Two-Period, Crossover Study to Compare Pharmacokinetic Properties of ARN-75039 Tablets With Excipients to Neat ARN-75039 in Hydroxypropyl Methylcellulose (HPMC) Capsules in Healthy Adult Participants Under Fed Conditions
Brief Title: A Comparison of the Pharmacokinetic Properties of ARN-75039 Tablets With Excipients to Neat ARN-75039 in Hydroxypropyl Methylcellulose (HPMC) Capsules in Healthy Adult Participants Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arisan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARN-75039-103
Record Dates: First submitted 2025-03-13; First posted 2025-04-04 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Lassa Virus Infection
MeSH Terms: conditions — Lassa Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): In Sequence 1, study participants are dosed with neat ARN-75039 in HPMC capsules (reference product) on Day 1 of Period 1. After a 7 day washout period, study participants are dosed with ARN-75039 with excipients in tablet form (comparator product) on Day 1 of Period 2.
  Interventions: Drug: ARN-75039
- Sequence 2 (Experimental): In Sequence 2, study participants are dosed with ARN-75039 with excipients in tablet form (comparator product) on Day 1 of Period 1. After a 7 day washout period, study participants are dosed with neat ARN-75039 in HPMC capsules (reference product).
  Interventions: Drug: ARN-75039

INTERVENTIONS:
Drug: ARN-75039 — An oral therapy for the treatment of Lassa infection

SUMMARY:
ARN-75039-103 is a comparative, randomized, single-dose, crossover study to assess the PK, safety, and tolerability of neat ARN-75039 in hydroxypropyl methylcellulose (HPMC) capsules against ARN 75039 with excipients in tablet form administered by the oral route in healthy adult participants. The safety assessments will include standard evaluations of vital signs, clinical laboratory values, and ECGs.

Participants will be admitted to the study site on the morning of Day -1, prior to Period 1 study drug administration, and will remain on site until Day 15. Upon confirmation of eligibility, participants will be randomized into the study on Day 1. Study drug administration will be performed on the first day of Periods 1 and 2 (Study Days 1 and 8, respectively) with a 7-day washout period between the two periods. Participants will receive the randomized study drug in the morning following a meal. A total of 16 participants will be randomized 1:1 to the following two sequences:

* Sequence 1:

  * Period 1: Neat ARN-75039 in HPMC capsules (reference product)
  * Period 2: ARN-75039 with excipients in tablet form (comparator)
* Sequence 2:

  * Period 1: ARN-75039 with excipients in tablet form (comparator)
  * Period 2: Neat ARN-75039 in HPMC capsules (reference product)

Participation in the study will be conducted in the following 5 defined periods:

* Screening Period: The Screening Period begins upon completion of the informed consent form (ICF). During this period, participants will undergo baseline assessments to determine eligibility for study participation. The Screening Period duration will be up to 21 days; it will end after all evaluations required to meet eligibility have been completed. If a participant meets all eligibility criteria, they will be offered enrollment into the study.
* Admission to Study Site: Participants will be admitted to the study site in the morning on the day prior to dosing of period 1 (Day -1). Participants that are eligible to participate in the study and are randomized into the study will remain at the study site until completion of the treatment period (Study Day 15).
* Treatment Period: This study consists of two treatment days separated by a 7-day washout period. The first treatment day will begin on Day 1 of Period 1 with administration of the first dose of study drug. The second treatment day will occur on the first day of Period 2 (Study Day 8). Following the dosing of the study drug on each treatment day, fifteen venous blood samples will be withdrawn via an indwelling cannula or by venipuncture at regular time intervals.
* End of Active Treatment (Day 15 Discharge Visit or Early Termination (ET) Visit): Upon successful completion of active treatment, participants will be discharged from the study site on Study Day 15. The Discharge Visit will include the completion of safety assessments, such as a physical examination, vitals, ECG recording, adverse event review, and clinical laboratory tests. Participants who complete both dosing days will be encouraged to complete all study visits.

Participants who do not complete all study visits or terminate from the study prior to Day 15 will be asked to complete the Early Termination Visit within 1 day after withdrawal from the study.

• Day 36 Telephone Follow Up Phone Call: Participants will be contacted by phone on Day 36-i.e., 28 days following the last study dose administered on Day 8. The purpose of this follow-up call is to assess for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

Participants meeting all the following criteria are eligible for study participation:

1. Is male or female, age 18 to 45 years, inclusive, at Screening.
2. Body mass index (BMI) between 18 and 35 kg/m2, inclusive, at Screening.
3. In good general health, determined by no clinically significant findings in the opinion of the Investigator from medical history, physical examination, 12-lead ECG, clinical laboratory findings, and vital signs at Screening and Day -1 or 1.
4. Hemoglobin, hematocrit, white blood cell count, absolute neutrophil count, and platelet count results within the laboratory reference range at Screening or without clinically significant abnormalities in the opinion of the Investigator; participants with Gilbert's disease with associated abnormalities of liver function tests are eligible for enrollment. Tests may be repeated at the discretion of the Investigator to confirm abnormalities.
5. Estimated glomerular filtration rate (eGFR) based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation of ≥ 80 mL/min/1.73 m2 at Screening.
6. Females of childbearing potential must practice effective contraception per national regulatory guidelines for clinical trials from Screening (see Section 5.6.2), throughout the study, and for 60 days after the last dose of study drug.
7. Females must have a negative pregnancy test at Screening and within 24 hours prior to dosing of study drug; for post-menopausal participants, a blood sample will also be tested for estradiol and follicle stimulating hormone (FSH) to confirm post-menopausal status based on reference laboratory ranges for post-menopausal status. Surgically sterile females are eligible; however, proof via medical records will be required.
8. Males must agree to not donate sperm and to use condom and spermicide in combination with any of the means of contraception for their female partners during sexual intercourse from the time of the first study drug administration and for 90 days following the last dose of study drug. Females must agree not to donate eggs from the time of the first study drug administration and for 60 days following the last dose of study drug.
9. Must be willing and able to comply with measures to avoid photosensitivity reactions (i.e., avoidance of outdoor sun exposure and tanning; consistent use of long sleeve shirts, long pants, hats, and sunglasses; consistent use of sun protection factor [SPF] 75 or greater sunscreen when outdoors) during the study treatment period.
10. Able to consume a standard meal (400-600 Calories) within 30 minutes.
11. Able to provide informed consent.
12. Willing and able to comply with this protocol and be available for the entire duration of the study.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for study participation:

1. Any clinically significant underlying illness in the opinion of the Investigator.
2. Poor venous access.
3. Prior exposure to ARN-75039.
4. History of drug or alcohol abuse within 1 year of Screening in the opinion of the investigator, or a positive test for drugs of abuse or alcohol at Screening or Day -1.
5. Use of any prescription or over-the-counter (OTC) medications, including food supplements, vitamins, herbal medications (e.g., St. John's wort), and cannabis, with the exception of contraceptive medications and as needed (prn) acetaminophen or paracetamol (not exceeding 2 grams/day) within 7 days prior to study drug administration and through the Day 15 Discharge visit.
6. Any female who is pregnant or breastfeeding, or any female who is planning to become pregnant during the study and safety follow-up period.
7. Currently enrolled in another investigational device or drug study, or less than 30 days or 5 half-lives of the prior investigational agent (whichever is longer) or plans to enroll in another investigational device or drug study during the course of this study.
8. Inability to ingest all capsules/tablets of a multi-capsule dose within 5 minutes of ingestion of the first capsule/tablet.
9. Positive serology for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) at Screening; participants with adequately treated HCV are eligible for enrollment.
10. Consumption of Seville oranges, grapefruit or grapefruit juice within 72 hours prior to Day 1 or during the study.
11. History of malignancy, except adequately treated basal cell carcinoma or in situ carcinoma of the uterine cervix.
12. Smoking cigarettes, cigars, cigarillos or E-cigarettes
13. Any reason or condition that, in the investigator's opinion, may compromise study participation, present a safety risk to the participant, or may confound the interpretation of the study results.
14. A QT duration corrected for heart rate by Fridericia's formula (QTcF) > 450 millisecond (msec) based on either single or averaged QTcF values of triplicate ECGs obtained over a 3-minute interval (at Screening).
15. Blood product (including plasma) donation within 30 days before Screening.
16. Unwilling to consume a breakfast on study drug administration days.
17. History of:

    * Structural abnormality of the GI tract or a disease or history of a condition that can affect GI motility.
    * Inflammatory bowel disease (even if treated and currently in remission).
    * Diverticulitis or any other chronic condition such as chronic pancreatitis, polycystic kidney disease, ovarian cysts, endometriosis, lactose intolerance that can be associated with abdominal pain or discomfort and could confound the assessments in this trial.
    * Chronic idiopathic diarrhea.
18. Formally diagnosed colonic inertia or conditions that can be associated with constipation: pseudo-obstruction, colonic inertia, megacolon, megarectum, bowel obstruction, descending perineum syndrome, solitary rectal ulcer syndrome, systemic sclerosis, lower tract evacuation disorders, functional outlet delay (e.g., rectal prolapse, anismus, etc.).
19. Current active peptic ulcer disease (i.e., disease that is not adequately treated or stable with therapy.)
20. Potential central nervous system cause of constipation (e.g., Parkinson's disease, spinal cord injury, and multiple sclerosis).
21. Participant currently has both unexplained and clinically significant alarm symptoms (lower GI bleeding [rectal bleeding or heme-positive stool], iron-deficiency anemia or any unexplained anemia, or weight loss) or systemic signs of infection or colitis.
22. History of chronic/generalized pruritus and/or skin rash of unknown origins.
23. Participants with diagnosed Type 1 or Type 2 diabetes, or with a fasting blood glucose value > 125 mg/dL during the screening period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
AUC0-t | 36 days
  Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration.
AUC0-24 | 36 days
  Area under the plasma concentration-time curve from time zero to 24 hours post-dose
AUC0-∞ | 36 days
  Area under plasma concentration-time curve from time zero to infinity
Cmax | 36 days
  Maximum observed plasma concentration
Cmin0-24 | 36 days
  Minimum observed plasma concentration from time zero to 24 hours post-dose
tmax | 36 days
  Time to reach Cmax
t1/2 | 36 days
  Half-life
CL/F | 36 days
  Apparent clearance after extravascular administration
Vz/F | 36 days
  o Apparent volume of distribution during the terminal phase after extravascular administration

SECONDARY OUTCOMES:
TEAEs | 36 days
  Type and frequency of treatment-emergent adverse events (TEAEs).
TESAEs | 36 days
  Type and frequency of treatment-emergent serious adverse events (TESAEs).
Greater than Grade 1 TEAEs | 36 days
  Type and frequency of study drug-related >Grade 1 TEAEs

CONTACTS AND LOCATIONS:
Overall Officials: Ken McCormack, PhD, Study Chair — Arisan Therapeutics
Locations (1):
- Frontage, Secaucus, New Jersey, United States